CLINICAL TRIAL: NCT04822584
Title: Evaluation of Effect and Tolerance of the Association of Baricitinib (4 mg) and Phototherapy Versus Phototherapy in Adults With Progressive Vitiligo: a Randomized, Double-blind, Prospective, Non-comparative Phase II Study.
Brief Title: Evaluation of Effect and Tolerance of the Association of Baricitinib and Phototherapy Versus Phototherapy in Adults With Progressive Vitiligo
Acronym: BARVIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2019/21
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Vitiligo
Keywords: vitiligo; phototherapy; baricitinib; randomized
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, non-comparative, phase II proof-of-concept trial involved patients with progressive vitiligo and uses one of the most common regimens in this phase of study. Assessment of the experimental treatment efficacy will be estimated only on the results obtained in the experimental treatment arm (baricitinib 4 mg/day + narrowband UVB TL01 arm).
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. To preserve the blinding of the study, a minimum number of sponsor personnel will see the randomization table and treatment assignments before the study is complete.
  All study assessments will be performed by study personnel who are blinded to the patient's treatment group.
  Except in clinical circumstances where unblinding is required, the patients, investigators, sponsor study team, and any personnel interacting directly with patients or investigative sites will remain blinded to baricitinib and placebo assignment until after completion of the Double-Blinded Treatment Period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phototherapy associated with active treatment (Experimental): Baricitinib 4 mg/day orally for 36 weeks + UVB TL01: 2 times a week during 24 weeks.
  (Phototherapy will be started 12 weeks after the beginning of baricitinib)
  Interventions: Drug: Baricitinib Oral Product
- Phototherapy associated with placebo (Placebo Comparator): Placebo once a day orally for 36 weeks + UVB TL01: 2 times a week during 24 weeks.
  (Phototherapy will be started 12 weeks after the beginning of placebo of baricitinib).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib Oral Product — Baricitinib 4 mg/day orally for 36 weeks
  Arms: Phototherapy associated with active treatment
Drug: Placebo — Placebo once a day orally for 36 weeks
  Arms: Phototherapy associated with placebo

SUMMARY:
The purpose of this phase 2 study is to evaluate the effect and the safety of the combination of Baricitinib in combination with phototherapy in adult participants with non-segmental progressive vitiligo.

DETAILED DESCRIPTION:
Treatment Strategy: Multicentric, parallel double blind randomized phase 2 prospective study comparing baricitinib (4mg/day) + narrowband UVB TL01 versus placebo + narrowband UVB TL01 Follow-up of the study: patients included in this study will start Baricitinib 3 months before starting narrowband UVB TL01. Phototherapy will be performed twice a week during 6 months. Follow-up visit will be done at week 12, 24, 36 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Subject: male or female aged ≥ 18 years and ≤ 75 years
* Diagnosis of non-segmental (symmetrical) vitiligo with a body surface area involved >5% excluding hands and feet
* Active non-segmental vitiligo is defined by:

  * Non-segmental vitiligo with new patches or extension of old lesions during the last 6 months AND
  * Presence of hypochromic aspect under Wood's lamp examination and/or perifollicular hypopigmentation under Wood's lamp examination.
* Able to read, understand, and give documented (electronic or paper signature) informed consent
* Registered in the French Social Security
* Agree to discontinue the use of the following excluded medications/treatments for at least 4 weeks prior to randomization (Visit 2) and throughout the study: systemic steroids, phototherapy, methotrexate, cyclosporine, mycophenolate mofetil, and azathioprine.
* Agree to discontinue the use of the following excluded medications for at least 2 weeks prior to randomization (Visit 2) and throughout the study:

  * TCS or topical immune modulators (e.g., tacrolimus or pimecrolimus)
  * Topical phosphodiesterase type 4 (PDE-4) inhibitor (crisaborole)
  * Topical JAK inhibitor (e.g., tofacitinib or ruxolitinib) and/or any other investigational topical treatments.
* Patient characteristics
* Are male or nonpregnant, nonbreastfeeding female patients, except:

  1. Male patients must agree to use 2 forms of birth control (1 must be highly effective, see below) while engaging in sexual intercourse with female partners of childbearing potential while enrolled in the study and for at least 4 weeks following the last dose of investigational product.
  2. Female patients of childbearing potential must agree to use 2 forms of birth control, when engaging in sexual intercourse with a male partner while enrolled in the study and for at least 4 weeks following the last dose of investigational product.

     The following birth control methods are considered acceptable (the patient should choose 2 to be used with their male partner, and 1 must be highly effective):
     * Highly effective birth control methods: oral, injectable, or implanted hormonal contraceptives (combined estrogen/progesterone or progesterone only, associated with inhibition of ovulation); intrauterine device or intrauterine system (e.g., progestin-releasing coil); or vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate).
     * Effective birth control methods: condom with a spermicidal foam, gel, film, cream, or suppository; occlusive cap (diaphragm or cervical/vault caps) with a spermicidal foam, gel, film, cream, or suppository; or oral hormonal contraceptives.
  3. Females of nonchildbearing potential are not required to use birth control and they are defined as:

     * Women ≥60 years of age or women who are congenitally sterile, or
     * Women ≥40 and <60 years of age who have had a cessation of menses for ≥12 months and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (≥40 mIU/mL or ≥40 IU/L), or women who are surgically sterile (i.e., have had a hysterectomy or bilateral oophorectomy or tubal ligation).
* Signed informed consent form (ICF)

Exclusion Criteria:

* Segmental or mixed vitiligo
* Patients that are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus) that would interfere with evaluations of the effect of study medication on vitiligo
* Patients who are currently experiencing a skin infection that requires treatment, or who are currently being treated with topical or systemic antibiotics.

Note: Patients may not be rescreened until at least 4 weeks after the date of their previous screen failure and at least 2 weeks after resolution of the infection.

* Patients that have any serious concomitant illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring. (e.g., unstable chronic asthma).
* Patients that have been treated with the following therapies:

  1. Monoclonal antibody (e.g., ustekinumab, omalizumab, dupilumab) for less than 5 half-lives prior to randomization.
  2. Received prior treatment with any oral JAK inhibitor (e.g., tofacitinib,ruxolitinib)
  3. Received any systemic corticosteroid administered within 4 weeks prior to planned randomization or are anticipated to require systemic corticosteroids during the study.
  4. Have had an intra-articular corticosteroid injection within 4 weeks prior to planned randomization.
  5. Have received more than 250 sessions of UV lights therapies.
* Patients that are largely or wholly incapacitated permitting little or no self-care, such as being bedridden.
* Patients that have uncontrolled arterial hypertension characterized by a repeated systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg in a seated position.
* Patients that have had any major surgery within 8 weeks prior to screening or that will require major surgery during the study that, in the opinion of the investigator, would pose an unacceptable risk to the patient.
* Patients that are immunocompromised and, in the opinion of the investigator, at an unacceptable risk for participating in the study.
* Patients that have experienced any of the following event within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Patients that have a history of recurrent (≥ 2) VTE or are considered at high risk of VTE as deemed by the investigator.
* Patients that have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
* Patients that have a history of lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for less than 5 years :

  1. Patients with cervical carcinoma in situ that has been resected with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study.
  2. Patients with basal cell or squamous epithelial skin cancers that have been completely resected with no evidence of recurrence for at least 3 years may participate in the study.
* Patients that have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection, including but not limited to the following:

Note: A recent viral upper respiratory tract infection or uncomplicatedurinary tract infection should not be considered clinically serious.

1. symptomatic herpes zoster infection within 12 weeks prior to screening.
2. history of disseminated/complicated herpes zoster (e.g., multidermatomal involvement, ophthalmic zoster, CNS involvement, or post-herpetic neuralgia).
3. symptomatic herpes simplex at the time of randomization.
4. active or chronic viral infection from hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
5. household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB.
6. evidence of active TB or have previously had evidence of active TB and did not receive appropriate and documented treatment.
7. clinically serious infection or received intravenous antibiotics for an infection, within the past 4 weeks of randomization.
8. any other active or recent infection within 4 weeks of randomization that, in the opinion of the investigator, would pose an unacceptable risk to the patient if participating in the study.

   * Patients that have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination).

Note: Patients eligible for herpes zoster vaccine, who have not received it prior to screening will be encouraged (per local guidelines) to do so prior to randomization; vaccination must occur >4 weeks prior to randomization and start of investigational product. Patients will be excluded if they were exposed to herpes zoster vaccination within 4 weeks of planned randomization.

Investigators should review the vaccination status of their patients and follow the local guidelines for vaccination of those ≥18 years of age with nonlive vaccines intended to prevent infectious disease prior to entering patients into the study

* Have a history of chronic alcohol abuse, IV drug abuse, or other illicit drug abuse within the 2 years prior to screening.
* Presence of significant uncontrolled neuropsychiatric disorder, are clinically judged by the investigator to be at risk for suicide.
* Have donated more than a single unit of blood within 4 weeks prior to screening or intend to donate blood during the course of the study.

Other non inclusion criteria:

* Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.
* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have participated within the last 30 days in a clinical study involving an investigational product. If the previous investigational product has a long half-life (2 weeks or longer), at least 3 months or 5 half-lives (whichever is longer) should be allowed between the end of the previous treatment and the inclusion.
* Have previously been randomized in this study or any other study investigating baricitinib.
* Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Diagnostic Assessments

* Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator, are clinically significant and indicate an unacceptable risk for the patient's participation in the study.
* Have evidence of active TB or latent TB:

  1. have evidence of active TB, defined in this study as the following:

     * Documented by a positive PPD test (≥5 mm induration between approximately 48 and 72 hours after application, regardless of vaccination history), medical history, clinical features, and abnormal chest x-ray at screening.
     * The QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. Patients are excluded from the study if the test is not negative and there is clinical evidence of active TB.

Exception: Patients with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT® TB test but must have a chest x-ray at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Score with Vitiligo Area Scoring Index (VASI) | week 36
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.

SECONDARY OUTCOMES:
Score with VASI score | week 12
  Change in percentage of repigmented Surface area 12 weeks after-inclusion, by using the VASI score at week 12.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
Score with VASI score | week 24
  Change in percentage of repigmented Surface area 24 weeks after-inclusion, by using the VASI score at week 24.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
Score with VASI score | week 48
  Change in percentage of repigmented Surface area 48 weeks after-inclusion, by using the VASI score at week 48.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
Evaluation of Face Vitiligo Aera Scoring Index (F-VASI) score | week 12
  Mean variation in percentage of Face Vitiligo Aera Scoring Index (F-VASI) score between baseline , week 12
Evaluation of Face Vitiligo Aera Scoring Index (F-VASI) score | week 24
  Mean variation in percentage of Face Vitiligo Aera Scoring Index (F-VASI) score between baseline , week 24
Evaluation of Face Vitiligo Aera Scoring Index (F-VASI) score | week 36
  Mean variation in percentage of Face Vitiligo Aera Scoring Index (F-VASI) score between baseline , week 36
Evaluation of Face Vitiligo Aera Scoring Index (F-VASI) score | week 48
  Mean variation in percentage of Face Vitiligo Aera Scoring Index (F-VASI) score between baseline , week 48
Number of Adverse Events (AE) and serious adverse events (SAE), as well as the proportion of discontinuation due to AEs and/or SAEs | week 36
  AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related, that occurs after a subject provides informed consent. Abnormal laboratory values or test results occurring after informed consent constitute AEs only if they induce clinical signs or symptoms, are considered clinically meaningful, require therapy, or require changes in the study drug.
Evaluation of score Vitiligo European Task Force (VETF) | Week 12
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score Vitiligo European Task Force (VETF) | Week 24
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score of the Vitiligo Extent Score (VES) | Week 36
  Variation in percentage of the Vitiligo Extent Score (VES). The VES score is used to assess the severity and extent of vitiligo. Using the VES calculator www.vitiligo-calculator.com, investigator choose the pictures that best represent the patient's skin lesions and then the percentage of depigmented area is calculated.
Evaluation of score of the Vitiligo Extent Score (VES) | Week 48
  Variation in percentage of the Vitiligo Extent Score (VES). The VES score is used to assess the severity and extent of vitiligo. Using the VES calculator www.vitiligo-calculator.com, investigator choose the pictures that best represent the patient's skin lesions and then the percentage of depigmented area is calculated.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 12
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 24
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 36
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 48
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Dermatology Life Quality Index (DLQI) | week 12
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) | week 24
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) | week 36
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) | week 48
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of the score of the Skindex 29 | Week 12
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Skindex 29 | Week 24
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Skindex 29 | Week 36
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Skindex 29 | Week 48
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | day 1
  Expression of IFN-α, TNF-α, IFN-γ, IL-4, IL-5, IL-12, IL-13, IL-15, IL-17, IL-22, IL-23, IL-33 CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, soluble HSP70.
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | week 12
  Expression of IFN-α, TNF-α, IFN-γ, IL-4, IL-5, IL-12, IL-13, IL-15, IL-17, IL-22, IL-23, IL-33 CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, soluble HSP70.
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | week 36
  Expression of IFN-α, TNF-α, IFN-γ, IL-4, IL-5, IL-12, IL-13, IL-15, IL-17, IL-22, IL-23, IL-33 CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, soluble HSP70.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Seneschal, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Service de Dermatologie - Hôpital Saint-André, Bordeaux
  - Service de dermatologie - Hôpital Henri Mondor - EA EpiDermE (Epidémiologie en Dermatologie et Evaluation des Thérapeutiques), Créteil
  - Centre Hospitalier Universitaire de Nice - Service de Dermatologie, Nice
  - Service de dermatologie Centre de Référence des Maladies Rares de la Peau et des muqueuses d'origine génétique - Hôpital Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seneschal J, Guyon M, Merhi R, Mazereeuw-Hautier J, Andreu N, Cazenave S, Ezzedine K, Passeron T, Boniface K. Combination of Baricitinib and Phototherapy in Adults With Active Vitiligo: A Randomized Clinical Trial. JAMA Dermatol. 2025 Apr 1;161(4):375-382. doi: 10.1001/jamadermatol.2024.5737. PMID 39841460